CLINICAL TRIAL: NCT00396123
Title: Effects Of Darbepoetin On Vascular Repair Mechanisms In Kidney Disease The DARBEPC Study
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Crystal A. Gadegbeku, Associate Professor of Internal Medicine, Nephrology, University of Michigan
Other Study IDs: HUM 7825
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Chronic Kidney Disease; Anemia
Keywords: Chronic Kidney Disease; Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Humans have cells in their blood stream called endothelial progenitor cells or EPCs. These are thought to be important in keeping blood vessels healthy. People with chronic kidney disease (CKD) have low numbers of these cells. People with cardiovascular (heart and blood vessel) disease also have low numbers. Patients with CKD have more cardiovascular disease then any other group.Erythropoietin is a hormone made by the kidneys. It is essential for making red blood cells and also activates EPCs. It is low in people with kidney disease.

As part of your regular medical care for correcting your low red blood cell count, you will be receiving a medication that acts like erythropoietin. It is called darbepoetin.

The purpose of this study is to see if darbepoetin treatment affects EPC numbers and function.

DETAILED DESCRIPTION:
The majority of patients with kidney disease, an estimated 20 million adults in the U.S., will die of cardiovascular disease. Further, the risk for cardiovascular events is 2-3 fold higher than in the general population and increases with the severity of renal impairment [1]. Reasons for this accelerated atherosclerotic process are unclear. Recent evidence suggests that endothelial progenitor cells (EPC) are critical to maintaining vascular integrity [2]. Patient populations with low circulating EPCs, including patients with kidney disease, have excess vascular disease burden. The hematopoietic cytokine, erythropoietin, is a key regulator of EPCs and is reduced in patients with kidney disease [3]. Therefore, we hypothesize that supplementation with the erythropoietin analog, darbepoetin, enhances EPC function leading to improvement in vascular repair mechanisms in patients with chronic (CKD).

To begin to explore this hypothesis, we will pursue the following specific aims.

1. Determine the effects of darbepoetin on EPC number in patients with anemia related to CKD
2. Determine the effects of darbepoetin on EPC function in patients with anemia related to CKD
3. Determine the effects of darbepoetin on proangiogenic factors in patients with anemia related to CKD

These studies will expand our understanding and potentially guide therapy aimed at reducing the excess cardiovascular disease burden in high risk populations.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in University of Michigan's Nephrology Anemia Clinic
* 18 years old or older
* Have kidney disease but are not on dialysis

Exclusion Criteria:

* Not enrolled in University of Michigan's Nephrology Anemia Clinic
* Less than 18 years of age
* Hematocrit that is less than 28.5%
* Currently participating in a clinical trial with an intervention
* Planning to change their tobacco use habits during the study period
* Have had dose changes of certain medications for cholesterol or diabetes within one month of study enrollment
* Are currently receiving:

  * darbepoetin
  * erythopoietin
  * medications to lower your immune system
* Have had problems within the last 3 months with:

  * Bleeding
  * Heart attack or stroke
  * Heart or blood vessel procedures
* Are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nephrology clinic
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2006-11; Primary Completion 2008-07-25 (Actual); Study Completion 2008-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal A Gadegbeku, MD, Principal Investigator — University of Michigan/Internal Medicine/Nephrology
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States